CLINICAL TRIAL: NCT02720471
Title: Local Analgesia Versus Local Peroperative Infiltration After Total Hip Replacement
Acronym: ALRIAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL15_0189
Record Dates: First submitted 2015-12-15; First posted 2016-03-28 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Total Hip Replacement
Keywords: local analgesia; total hip replacement; local infiltrations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Locoregional anesthesia (Active Comparator): Classical locoregional analgesia by ultrasound guidance by blocks of the femoral and cutaneous nerves side of the thigh will be performed in patients of this arm
  Interventions: Drug: Locoregional anesthesia
- Peroperative infiltration (Experimental): Peroperative infiltration of local anesthetics (IAL) will be performed in patients of this arm
  Interventions: Drug: peroperative infiltration of local anesthetics

INTERVENTIONS:
Drug: Locoregional anesthesia — classical analgesia by ultrasound guidance by blocks of the femoral and cutaneous nerves side of the thigh
  Arms: Locoregional anesthesia
Drug: peroperative infiltration of local anesthetics — peroperative infiltration of local anesthetics
  Arms: Peroperative infiltration

SUMMARY:
Clinical study, comparative, prospective, interventional, randomized, single-center, single-blind The fast resumption of the walking after surgery of total prosthesis of hip (PTH) requires an effective analgesia from the immediate post-operative period. In France, whatever is the peroperative anesthesia, the analgesic reference technique is a locoregional anesthesia (ALR) ultrasound guidance by blocks of the femoral and cutaneous nerves side of the thigh. In the Anglo-Saxon countries, in particular in Australia and in the United States, the techniques of peroperative infiltration of local anesthetics (IAL) by the surgeon supplanted the techniques of traditional ALR. However, no French study compares the IAL with the conventional ALR with a rigorous methodology. Our occasional practice of IAL suggests us that it is more effective in terms of post-operative analgesia with Analog Visual Scales decreased (EVA) and a lesser consumption of morphine. Furthermore, the resumption of the upright posture in bipedal support as well as the resumption of the walking would be earlier.

The main objective is to show that the post-operative analgesia by local peroperative infiltration is superior to that obtained by locoregional anesthesia (ALR by femoral block associated with a side cutaneous block of the thigh) after the surgery of total prosthesis of hip, with decrease of the consumption of morphine within first 72 post-operative hours.

The secondary objectives are to compare the Analog Visual Scales of pain (EVA) with the rest and with the mobilization during various times (in post-surgery care room, then at H4, H8, H12, H24, H48, H72), the period between the end of intervention (out of the operating room) and the first support by the upright posture in bipedal support), the period between the end of intervention and the resumption of the walk, the satisfaction of the patients at the exit of the hospital, the duration of hospitalization after the surgical operation and the possible unwanted events (systematic toxicity of the local anesthetics, the infection of prosthesis, disease thromboembolic venous) during the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > or = 18 years old
* Surgery for total hip replacement (THR)
* Unilateral THR
* First THR
* THR planned because of a degenerative disease or after a traumatism
* Whatever the technique of anesthesia (general anesthesia or intra thecal anesthesia)
* Whatever the surgery technique/surgical approach
* Patient with a social security protection
* Patient not under juridic protection
* Agreement for the study signed by the patient himself or, if he is not able to sign, by his trusted person.

Exclusion Criteria:

* Patient Refusal
* Second hip replacement
* Pregnancy or breastfeeding
* Porphyria
* Risks to have methemoglobinemia (G6PD deficit, hemoglobin disease)
* BMI> 40 kg/m2 ou < 18 kg/m2
* Allergy to any of the drugs used in this study
* Contraindication to any of the technic used in this study
* Factors wich could influence the perception of pain (depression, dementia, psychiatric illness, neurologic disease with sensitivity troubles)
* Usual consumption of opioids
* Systemic or articular infection
* Participation to an other research that could interfere in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-09-14; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Quantity of morphine consumed | 72 hours after surgery
  Morphine consumption will be measured within the 72 hours following surgery

SECONDARY OUTCOMES:
Pain at rest | 72 hours after surgery
  Visual analogic pain scale (EVA) will be used to evaluate patient's pain at rest within the 72 hours following surgery
Pain while moving | 72 hours after surgery
  Visual analogic pain scale (EVA) will be used to evaluate patient's pain while moving within the 72 hours following surgery
Time between intervention and first support by the upright posture in bipedal station. | From date of surgery until the date of first documented resumption of walk, assessed up to 20 days after surgery
  Period between the end of intervention (out of the operating room) and the first support by the upright posture in bipedal station.
Time between intervention and resumption of the walk | From date of surgery until the date of first documented resumption of walk, assessed up to 20 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot - Département d'anesthésie réanimation, Lyon, France